CLINICAL TRIAL: NCT05917444
Title: Managing Breast Cancer Treatment: Dyad's Perspectives on Treatment Decision, Financial and Family Burden.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 202301195RINB
Record Dates: First submitted 2023-03-31; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; financial toxicity; Financial and Family Burden
MeSH Terms: conditions — Breast Neoplasms; Financial Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to understand the financial burden and treatment decisions, based on both of patient's and family's perspectives in breast cancer patients who receive systemic chemotherapy, targeted therapy or immuno-therapy and their family caregivers .

DETAILED DESCRIPTION:
This study utilizes a cross-sectional survey and qualitative research design. Data collection includes questionnaire surveys and recorded qualitative interviews. A total of 224 patients or family members who meet the criteria will be invited to participate in the study at oncology units and outpatient clinics. Among them, 30 subjects, either patients or family caregivers will be invited to explore their experience on and concerns about financial burden and treatment decision making as facing breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer

  1. Patients with newly diagnosed or recurrent breast cancer who require chemotherapy or targeted immunotherapy as recommended by their physicians
  2. Age 20 to 70
  3. Within 0.5 to 3 years of newly diagnosed or recurrent breast cancer
  4. Ability to perform housework or wage employment before cancer
  5. Those whose cognitive function is sufficient to read newspaper news and answer questionnaires
* breast cancer family

  1. Patient has been 0.5 to 3 years since the first diagnosis or recurrence of breast cancer and the doctor recommends chemotherapy or targeted immunotherapy
  2. Patient's self-reported family members who are involved in the patient's physical, social, or medical caregivers with cancer
  3. Age 20 to 65
  4. Able to perform housework or wage workers
  5. Those whose cognitive function is sufficient to read newspaper news and answer questionnaires

Exclusion Criteria:

* breast cancer

  1. Patients who were disabled before suffering from cancer
  2. only undergoing surgery or hormone therapy
* breast cancer family

  1. Persons with physical, mental and social disabilities
  2. Family members who are not involved in the patient's physical, social, or medical care for cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have diagnosed breast cancer and their family.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Chinese version of the short form 36 health survey questionnaire (SF-36) | within the past month
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
FACT-COST(COmprehensive Score for financial Toxicity) | Past 7 days
  instrument that assesses the degree of financial distress experienced by cancer patient,12-item COST-PROM the terms used to describe feelings about financial condition have been numerous, including perceived economic well being,personal financial wellness, financial satisfaction, perceived income adequacy, financial stress, debt stress, economic strain, and economic distress.Using the Likert five-point scale, the scores represent the following: 0 indicates 'completely absent,' 1 indicates 'very few,' 2 indicates 'few,' 3 indicates 'some,' and 4 indicates 'very many.' Higher scores indicate better economic conditions
M. D. Anderson Symptom Inventory | within 24 hours
  The first part of the MDASI consists of 13 single-item measures of symptom intensity, including fatigue, sleep disturbance, pain, drowsiness, poor appetite, nausea, vomiting, shortness of breath, numbness, difficulty remembering, dry mouth, distress, and sadness. Each symptom item is rated on a scale of 0 (not al all) to 10 (as bad as you can imagine). The second part of the MDASI assesses the extent to which symptoms interfere with general activities, mood, normal work, relations with other people, walking, and enjoyment of life. Each of the six interference items is rated on a scale of 0 (does not interfere) to 10 (completely interferes). A symptom severity composite score (average of the 13 symptom items) and an interference composite score (average of the six interference items) were computed.
Cancer Behavior Inventory-Brief | Past 7 days
  12-item measure of self-efficacy for coping, including:(1) Maintenance of Activity and Independence; (2) Coping with Treatment-Related Side Effects; (3) Accepting Cancer/Maintaining Positive Attitude; (4) Seeking and Understanding Medical Information; (5) Affective Regulation; (6) Seeking Support; and (7) Stress Management for Medical Appointments. Likert-type scale that ranged from 1 (not at all confident) to 9 (totally confident), reflecting the degree of confidence the patient has that he or she can perform that particular coping behavior.
Decisional Regret Scale | Past 7 days
  The Decision Regret Scale measures the level of regret that patients have regarding their overall cancer treatment. It consists of five items that assess feelings related to the rightness or wrongness of the decision, the harm caused, and whether they would make the same decision again after surgery. It is scored using a 5-point Likert scale, with higher scores indicating a greater level of regret.
Financial and Work ability Index | Past a month
  The self-administered questionnaire consists of 7 items, including aspects such as physical and mental ability, cognitive function, and health status of the worker. The scores of each item are summed up, resulting in a total score ranging from 7 to 49. A higher score indicates better work ability. The work ability is assessed based on the total score

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, Principal Investigator — National Taiwan University Hospital; Shiuyu C. LEe, Principal Investigator — National Taipei University of Nursing and Health Science
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan